CLINICAL TRIAL: NCT05504642
Title: Nivolumab and Ipilimumab for Chemo-radio-immunotherapy Followed by Maintenance Therapy With Nivolumab and Ipilimumab for Primary Treatment in Locally Advanced Cervical Cancer Patients
Brief Title: Chemo-radio-immunotherapy With Nivolumab and Ipilimumab Treatment in Locally Advanced Cervical Cancer Patients
Acronym: CERAD-IMMUNE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped before submission for funding reasons
Sponsor: Universitätsklinikum Köln (Other)
Collaborators: ZKS Köln (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-4513
Record Dates: First submitted 2022-03-01; First posted 2022-08-17 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Cervical Cancer ≥ FIGO IIB and or Lymph Node Metastases
Keywords: cervical cancer; lymph node metastases; FIGO IIB
MeSH Terms: conditions — Lymphatic Metastasis; Uterine Cervical Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Open-label, single-arm, monocenter phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study medication (Experimental): All eligible patients will receive study medication:
  * Pre-Chemo-radio-immunotherapy Treatment for two weeks before start of Chemo-radio-immunotherapy
  * Concurrent Chemo-radio-immunotherapy (week 1-7)
  * Maintenance Treatment (six months) after Chemo-radio-immunotherapy
  Interventions: Drug: Pre-Chemo-radio-immunotherapy Treatment (Nivolumab/Ipilimumab); Drug: Concurrent Chemo-radio-immunotherapy (Nivolumab/Ipilimumab); Procedure: Maintenance Treatment (Nivolumab/Ipilimumab)

INTERVENTIONS:
Drug: Pre-Chemo-radio-immunotherapy Treatment (Nivolumab/Ipilimumab) — Two weeks before start of Chemo-radio-immunotherapy one administration of Nivolumab 3 mg/kg and Ipilimumab 1 mg/kg IV over 30 minutes, with a 30 minute break between Nivolumab and Ipilimumab.
Drug: Concurrent Chemo-radio-immunotherapy (Nivolumab/Ipilimumab) — In week 1-7, standard administration of concurrent Cisplatin mono 40mg/m2 body surface area d1, 8, 15, 22, 29 (Monday of each treatment week) during radiotherapy. Simultaneous application of Nivolumab 3mg/kg week 1, 3, 5, 7 (on Thursday) and Ipilimumab 1mg/kg in week 5 (on Thursday).
Procedure: Maintenance Treatment (Nivolumab/Ipilimumab) — For six months after Chemo-radio-immunotherapy, Nivolumab 3mg/kg every two weeks x12 (week +2, +4, +6, +8, +10, +12, +14, +16, +18, +20, +22, +24 (twelve applications), each application over 30 minutes and Ipilimumab every six weeks x4 (week +6,+12, +18, +24).

SUMMARY:
The purpose of this study is to use Chemo-radio-immunotherapy and maintenance therapy with Nivolumab and Ipilimumab in order to achieve improved outcome in patients with locally advanced cervical cancer.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all eligible patients giving written informed consent will undergo a Pre-Chemo-radio-immunotherapy Treatment with Nivolumab and Ipilimumab for 2 weeks. In the following week 1-7, concurrent Chemo-radio-Immunotherapy will consist of standard administration of concurrent Cisplatin mono during radiotherapy, with simultaneous application of Nivolumab and Ipilimumab according to trial protocol. This is followed by Maintenance Treatment for 6 months with Nivolumab and Ipilimumab according to trial protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Fully-informed written consent.
2. Females ≥ 18 years of age
3. Histologically confirmed squamous cell, adeno- adenosquamous carcinoma of the cervix uteri. Surgical staging prior to treatement is optional.
4. FIGO stage ≥ IIB and/or histologically confirmed pelvic lymph node metastases.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
6. Adequate bone marrow, hepatic and renal function including the following:

   * Haemoglobin ≥ 9.0 g/dL, absolute neutrophil count ≥ 1,500 /µL, platelets ≥100,000 /µL;
   * Total bilirubin ≤ 1.5 x upper normal limit; (except subjects with Gilbert Syndrome who can have total bilirubin < 3.0 mg/dL);
   * AST (SGOT), ALT (SGPT) ≤ 3 x upper normal limit;
   * International normalized ratio (INR) ≤ 1.25;
   * Creatinine ≤ 1.5 x upper normal limit OR measured or calculated creatinine clearance (according to Cockcroft-Gault) ≥40 mL/min for participant with creatinine levels >1.5 × institutional ULN (GFR can also be used in place of creatinine or CrCl)
7. Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial. Women must not be breastfeeding.
8. The patient is willing and able to comply with the protocol for the duration of the study, including hospital visits for treatment and scheduled follow-up visits and examinations.
9. WOCBP must agree to follow instructions for method(s) of contraception for the treatment time and 5 months after.

Exclusion Criteria:

1. Previous systemic therapy in the first-line setting.
2. Patients with neuroendocrine (small cell or large cell) tumors or mixed neuroendocrine histology.
3. Patients with histologically confirmed para-aortic lymph node metastases.
4. Prior organ allograft or allogeneic bone marrow transplantation.
5. Local therapies ongoing or completed <4 weeks prior to the baseline scan.
6. Thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months prior to the first dose of study drug with the exception of thrombosis of a segmental portal vein.
7. Prior, systemic anti-cancer chemotherapy, radiotherapy administered <4 weeks prior to study entry, endocrine- or immunotherapy or use of other investigational agents.
8. Major surgery within 4 weeks of starting the study. Patients must have recovered from effects of major surgery.
9. Malignancies other than disease under study within 5 years prior to inclusion, with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year OS rate >90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent)
10. Any serious or uncontrolled medical disorder or active infection that, in the opinion of the investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the subject to receive study drug.
11. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or compliance with the study protocol.
12. Subjects with a history of or current CNS metastases. A scan to confirm the absence of brain metastases is not required. Patients with unknown CNS metastatic status and any clinical signs indicative of CNS metastases are eligible if CNS metastases are excluded using CT and/or MRI scans.
13. Pregnant or breast-feeding women.
14. Any positive test result for hepatitis B virus (e.g. surface antigen [HBV sAg, Australia antigen] positive) or hepatitis C virus (Hepatic C antibody [anti-HCV] positive, except if HCV-RNA negative.
15. Immunocompromised patients, e.g. patients with positive testing for HIV at screening visit or those under corticoid medication or immunosuppressive drugs (e.g. methotrexate).
16. Subjects with active, known, or suspected autoimmune disease. Subjects with Type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll. For any cases of uncertainty, it is recommended that the coordinating investigator be consulted prior to signing informed consent.
17. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
18. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
19. Non-resolved (> Grade 1 (NCI CTCAE version 5) toxicities attributed to prior anti-cancer therapy other than hearing loss, alopecia and fatigue
20. > Grade 1 peripheral neuropathy according to CTCAE version 5.
21. History of allergy or hypersensitivity to study drugs or any constituent of the products
22. Patient is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.23.Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG.24.Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From Baseline to 2 years
  Tumor response assessed by MRI Pelvic according to resist
The adverse events according to NCI-CTCAE v5.0 | From the time of signed informed consent until 100 days after the last study drug administration
  Safety and tolerability (according to NCI-CTCAE v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Simone Marnitz, Prof., Principal Investigator — Department of Radiation Oncology, University Hospital of Cologne